CLINICAL TRIAL: NCT04327024
Title: A Phase 2, Multicentre, Double-Blind, Placebo and Active Control Efficacy and Safety Study to Evaluate Verinurad Combined With Allopurinol in Heart Failure With Preserved Ejection Fraction
Brief Title: Study of Verinurad in Heart Failure With Preserved Ejection Fraction
Acronym: AMETHYST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5496C00005; 2019-004862-16 (EudraCT Number)
Record Dates: First submitted 2020-03-13; First posted 2020-03-30 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: Phase 2,; Double-Blind,; Placebo and Active Control,; Verinurad,; Allopurinol,; HFpEF,; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — verinurad; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Verinurad 12 + allopurinol (Experimental): Dose [mg] verinurad/allopurinol:
  Step 1 - titration_3/100 Step 2 - titration_7.5/200 Step 3 - target dose 12/300
  Interventions: Drug: Verinurad; Drug: Allopurinol
- Allopurinol alone (Experimental): Dose [mg] verinurad/allopurinol:
  Step 1 - titration_0/100 Step 2 - titration_0/200 Step 3 - target dose 0/300
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Placebo [mg] in 3 steps 0/0
  Interventions: Drug: Placebo for verinurad; Drug: Placebo for allopurinol

INTERVENTIONS:
Drug: Verinurad — The treatment will be titrated in 3 steps for target low dose (3 mg), intermediate dose (7.5 mg) and high dose (12mg) of verinurad.
  Drug: Allopurinol The treatment will be titrated in 3 steps. Low dose (100mg), intermediate (200mg) and high dose (300mg) of allopurinol.
  Other Names: verinurad titration 3 - 7.5 - 12mg; allopurinol titration 100 - 200 - 300 mg
  Arms: Verinurad 12 + allopurinol
Drug: Allopurinol — Study treatments will be titrated in 3 steps: Low dose (100mg), intermediate (200mg) and high dose (300mg) of allopurinol
  Other Names: allopurinol titration 100 - 200 - 300 mg
  Arms: Allopurinol alone; Verinurad 12 + allopurinol
Drug: Placebo for verinurad — Matching Capsule
  Other Names: Placebo
  Arms: Placebo
Drug: Placebo for allopurinol — Matching tablet
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
International, Multicenter, Double-Blind, Placebo and Active Control Efficacy and Safety Study to Evaluate Verinurad combined with Allopurinol in Heart Failure with Preserved Ejection Fraction

DETAILED DESCRIPTION:
Evidence shows independent associations between hyperuricaemia and the risk of cardio-renal conditions, including heart failure (HF). Serum uric acid (sUA) is also a strong prognostic factor and correlates with other markers of poor prognosis in HF patients with preserved ejection fraction (HFpEF), and an estimated 1/2-2/3 of HFpEF patients have hyperuricaemia. HFpEF is a microvascular disease likely partly driven by endothelial dysfunction and inflammation in coronary vessel walls. Uric acid crystals have been identified in coronary vessel walls in some hyperuricaemic patients.

Uric acid transporter 1 (URAT1) is responsible for reabsorption of uric acid (UA) in the proximal tubule. Inhibition of URAT1 results in increased urinary excretion of UA and lowering of uric acid in the blood. Verinurad is a novel URAT1 inhibitor in Phase 2 development for chronic kidney disease (CKD) and HF. Verinurad combined with the xanthine oxidase (XO) inhibitors (XOI) febuxostat or allopurinol has been shown to lower sUA in patients with recurrent gout in Phase 2 studies by up to approximately 80%.

The primary objective of this Phase 2 study is to assess the effect of a combination of verinurad and allopurinol on exercise capacity in patients with HFpEF.

The secondary objectives are to assess effect of combination of verinurad and allopurinol in comparison to allopurinol monotheraphy on excercise capacity dwhich will be measured in peak VO2 as well as effect of verinurad and allopurinol compared to placebo and to allopurinol monotheraphy on Kansas City cardiomyopathy questionnaire (KCCQ)-total symptom score (TSS). A sub-study aims to investigate the relationship between UA crystals and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 40 years of age at the time of signing the ICF
* Patients with hyperuricaemia defined as sUA level of > 6 mg/dL.
* Patients with documented diagnosis of symptomatic HFpEF according to all of the following criteria:

  1. Have NYHA functional class II-III at enrolment
  2. Have medical history of typical symptoms/signs of HF > 6 weeks before enrolment
  3. LVEF ≥ 45%
  4. NT-proBNP ≥ 125 pg/mL (≥ 14.75 pmol/L) at Visit 1 for patients without ongoing atrial fibrillation/flutter.
* Patients able to exercise to near exhaustion during a CPET as exhibited by RER

  ≥ 1.05 during CPET conducted during screening. If patient does not achieve RER ≥ 1.05 the CPET may be repeated once, at least 48 hours but less than 2 weeks (but before randomisation) after the initial test; in such cases the second test will serve as baseline.
* Male or female

Exclusion Criteria:

* eGFR < 30ml/min/1.73m2 (based on CKD-EPI formula)
* Presence of any condition that precludes exercise testing
* Known history of a documented LVEF < 40%
* Probable alternative or concomitant diagnoses which in the opinion of the Investigator could account for the patient's HF symptoms and signs (eg, anaemia, hypothyroidism)
* Known carrier of the Human Leukocyte Antigen-B (HLA-B) *58:01 allele: HLA-B

  *58:01 genotyping is mandatory prior to randomization for all patients.
* Patients diagnosed with tumor lysis syndrome or Lesch-Nyhan syndrome
* Patients who are severely physically or mentally incapacitated and who in the opinion of investigator are unable to perform the patients' tasks associated with the protocol
* Presence of any condition which, in the opinion of the investigator, places the patient at undue risk or potentially jeopardises the quality of the data to be generated
* Current acute decompensated HF or hospitalisation due to decompensated HF < 4 weeks prior to enrolment
* Myocardial infarction, unstable angina, coronary revascularisation (percutaneous coronary intervention or coronary artery bypass grafting), ablation of atrial flutter/fibrillation, valve repair/replacement, implantation of a cardiac resynchronisation therapy device, stroke or transient ischemic attack within 6 months prior to enrolment.
* Planned coronary revascularisation, ablation of atrial flutter/fibrillation and/or valve repair/replacement
* Atrial fibrillation with persistent resting heart rate > 110 beats per minute.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalane Kitzman, MD, Principal Investigator — 1326 Riverview Road Ext Lexington, NC 27292-1764 USA
Locations (44):
- United States (8):
  - Research Site, Granada Hills, California
  - Research Site, Northridge, California
  - Research Site, Torrance, California
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Norfolk, Virginia
- Argentina (3):
  - Research Site, CABA
  - Research Site, Mar del Plata
  - Research Site, Rosario
- Australia (4):
  - Research Site, Bedford Park
  - Research Site, Chermside
  - Research Site, Geelong
  - Research Site, Milton
- Austria (2):
  - Research Site, Graz
  - Research Site, Vienna
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Research Site, Québec, Quebec, Canada
- Germany (5):
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Göttingen
  - Research Site, Regensburg
  - Research Site, Würzburg
- Research Site, Querétaro, Mexico
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Chrzanów
  - Research Site, Lublin
  - Research Site, Tychy
  - Research Site, Warsaw
- Russia (5):
  - Research Site, Aramil
  - Research Site, Kemerovo
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
- Slovakia (4):
  - Research Site, Brezno
  - Research Site, Lučenec
  - Research Site, Prešov
  - Research Site, Svidník
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Gangwon-do
  - Research Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Kitzman DW, Voors AA, Mentz RJ, Lewis GD, Perl S, Myte R, Kaguthi G, Sjostrom CD, Kallgren C, Shah SJ. Verinurad Plus Allopurinol for Heart Failure With Preserved Ejection Fraction: The AMETHYST Randomized Clinical Trial. JAMA Cardiol. 2024 Oct 1;9(10):892-900. doi: 10.1001/jamacardio.2024.2435. PMID 39141378
- See also: Clinical Study Protocol Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5496C00005&attachmentIdentifier=fce5ac49-abba-45d6-97e6-9c743db21176&fileName=Clinical_Study_Protocol_redacted.pdf&versionIdentifier=
- See also: CSR_synopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5496C00005&attachmentIdentifier=99f91757-f330-4480-b3fa-db052dbed5ca&fileName=Clinical_Study_Report_synopsis_redacted.pdf&versionIdentifier=
- See also: Statistical Analysis Plan-redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5496C00005&attachmentIdentifier=d1b3f66a-e0b3-4c29-bd75-cbabdfcc4f19&fileName=Statistical_Analysis_Plan-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 475 subjects were screened between May 19, 2020, and July 16, 2021, at 59 sites in 12 different countries. Of those screened, 159 were randomized into the study and received treatment, 53 in each arm of the study.
Pre-assignment Details: Subjects who met all the of inclusion criteria and none of the exclusion criteria were randomized to a study treatment. Study treatment was titrated over 8 weeks. Colchicine prophylaxis was given during the titration period and during the first 4 weeks of treatment at target dose (12 weeks total) and was distributed as available, currently 500 μg within the European Union (EU) and 600 μg within the United States (US).
Groups:
- Verinurad + Allopurinol: 12 mg verinurad + 300 mg allopurinol
- Allopurinol: 300 mg Allopurinol
- Placebo: 0 mg placebo
Period: Overall Study
Arm/Group | Verinurad + Allopurinol | Allopurinol | Placebo
Started | 53 | 53 | 53
Completed | 51 | 49 | 50
Not Completed | 2 | 4 | 3
Not completed — Death | 1 | 2 | 1
Not completed — Non-compliance with study drug | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set includes all subjects who have been randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Verinurad + Allopurinol | Allopurinol | Placebo | Total
Number analyzed (Participants) | 53 | 53 | 53 | 159
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.6 (9.04) | 70.6 (6.98) | 67.5 (9.77) | 69.2 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 16 | 56
  Male | 32 | 34 | 37 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 4 | 13
  Not Hispanic or Latino | 50 | 47 | 49 | 146
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 46 | 46 | 48 | 140
  Black or African American | 0 | 3 | 1 | 4
  Asian | 7 | 3 | 4 | 14
  Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at Week 32 in Peak V02 Consumption in Verinurad + Allopurinol Compared to Placebo (ANCOVA Model)
Description: Mean change from baseline in peak VO2 at Week 32 between the treatment groups was compared using change from baseline (i.e., week 32 value - baseline value) as the dependent variable, treatment as the independent variable and baseline peak VO2 included as covariate.
  H0: Difference in mean change from baseline in peak VO2 (verinurad + allopurinol vs placebo) = 0 Ha: Difference in mean change from baseline in peak VO2 (verinurad + allopurinol vs placebo) ≠ 0
  A hierarchical test sequence was used for the confirmatory analysis of the primary and secondary objectives in order to address the issue of multiple testing and control the Type I error rate at an overall two-sided 0.05 level.
  Since this was the first test in the hierarchical test sequence and endpoint was not rejected at a two-sided 0.05 level, the testing sequence did not continue.
Time Frame: From baseline to Week 32
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg/min
Arm/Group | Verinurad + Allopurinol | Placebo
Number analyzed (Participants) | 53 | 53
mL/kg/min | 0.27 [-0.56 to 1.10] | 0.37 [-0.45 to 1.19]
Statistical Analysis 1: Comparison: Verinurad + Allopurinol vs Placebo; Test type: Other; p = 0.862, ANCOVA; Model included change from baseline as the dependent variable, treatment as the independent variable and baseline peak VO2 as covariate; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-1.28 to 1.08]

2. Secondary Outcome: Change From Baseline at Week 32 in Peak V02 Consumption in Verinurad+ Allopurinol Compared to Allopurinol Monotherapy (ANCOVA Model)
Description: Mean change from baseline in peak VO2 at Week 32 between the treatment groups was compared using change from baseline (i.e., week 32 value - baseline value) as the dependent variable, treatment as the independent variable and baseline peak VO2 included as covariate.
  H0: Difference in mean change from baseline in peak VO2 (verinurad + allopurinol vs allopurinol) = 0 Ha: Difference in mean change from baseline in peak VO2 (verinurad + allopurinol vs allopurinol) ≠ 0
  A hierarchical test sequence was used for the confirmatory analysis of the primary and secondary objectives in order to address the issue of multiple testing and control the Type I error rate at an overall two-sided 0.05 level.
Time Frame: From baseline to Week 32
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/Kg/min
Groups:
- Allopurinol Monotherapy: 300 mg allpurinol
Arm/Group | Verinurad + Allopurinol | Allopurinol Monotherapy
Number analyzed (Participants) | 53 | 53
mL/Kg/min | 0.27 [-0.56 to 1.10] | -0.17 [-1.03 to 0.69]
Statistical Analysis 1: Comparison: Verinurad + Allopurinol vs Allopurinol Monotherapy; Test type: Other; p = 0.472, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.76 to 1.64]

3. Secondary Outcome: Change From Baseline at Week 32 in KCCQ-TSS in Verinurad+ Allopurinol Compared to Placebo (MMRM)
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item assessment that measures the patient's perception of their health status, which includes heart failure-related symptoms (frequency, burden, recent change), impact on physical and social function, self-efficacy and knowledge, and how the patient's heart failure affects their quality of life. The Total Symptom Score (TSS) averages the frequency domain and the symptom burden domain subscales, which each range from 0 to 100. The TSS ranges from 0-100 (higher scores = better health status).
  Mean change from baseline in KCCQ-TSS at Week 32 between the treatment groups was compared using MMRM analysis, with change from baseline (i.e., week 32 value - baseline value) as the dependent variable, treatment as the independent variable and visit, visit by treatment, and baseline KCCQ-TSS included as covariates.
  The number analyzed at each timepoint represents the number of subjects with data at each visit.
Time Frame: From baseline to Week 22 and Week 32
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Verinurad + Allopurinol | Placebo
Number analyzed (Participants) | 53 | 53
Scores on a scale
  Week 22: number analyzed (Participants) | 51 | 48
  Week 22 | 0.50 [-4.08 to 5.08] | 3.55 [-1.29 to 8.39]
  Week 32: number analyzed (Participants) | 51 | 48
  Week 32 | 4.31 [0.28 to 8.33] | 1.16 [-3.02 to 5.34]
Statistical Analysis 1: Comparison: Verinurad + Allopurinol vs Placebo; H0: Difference in mean change from baseline in KCCQ-TSS (verinurad + allopurinol vs placebo) = 0 Ha: Difference in mean change from baseline in KCCQ-TSS (verinurad + allopurinol vs placebo) ≠ 0 A hierarchical test sequence was used for the confirmatory analysis of the primary and secondary objectives in order to address the issue of multiple testing and control the Type I error rate at an overall two-sided 0.05 level; Test type: Other; p = 0.287, Mixed Models Analysis; Model included treatment as the independent variable and visit, visit by treatment, and baseline KCCQ-TSS as covariates; Mean Difference (Final Values) = 3.15, 95% CI 2-sided [-2.65 to 8.94]

4. Secondary Outcome: Change From Baseline at Week 32 in KCCQ-TSS in Verinurad+ Allopurinol Compared to Allopurinol Monotherapy (MMRM)
Description: as for outcome 3
Time Frame: From baseline to Week 22 and Week 32
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- Allopurinol Monotherapy: 300 mg allopurinol
Arm/Group | Verinurad + Allopurinol | Allopurinol Monotherapy
Number analyzed (Participants) | 53 | 53
Scores on a scale
  Week 22: number analyzed (Participants) | 51 | 50
  Week 22 | 0.50 [-4.08 to 5.08] | 2.85 [-1.91 to 7.62]
  Week 32: number analyzed (Participants) | 51 | 50
  Week 32 | 4.31 [0.28 to 8.33] | 4.45 [0.34 to 8.57]
Statistical Analysis 1: Comparison: Verinurad + Allopurinol vs Allopurinol Monotherapy; H0: Difference in mean change from baseline in KCCQ-TSS (verinurad + allopurinol vs allopurinol) = 0 Ha: Difference in mean change from baseline in KCCQ-TSS (verinurad + allopurinol vs allopurinol) ≠ 0 A hierarchical test sequence was used for the confirmatory analysis of the primary and secondary objectives in order to address the issue of multiple testing and control the Type I error rate at an overall two-sided 0.05 level; Test type: Other; p = 0.960, Mixed Models Analysis; Model included treatment as the independent variable and visit, visit by treatment, and baseline KCCQ-TSS as covariates; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-5.90 to 5.61]

ADVERSE EVENTS:
Time Frame: Adverse events were collected with onset date on or after first dose and up to the end of the study (week 36). Serious adverse events were collected with onset date on or after the signing of the informed consent form and up to the end of the study (week 36).
Description: All adverse events reported are treatment emergent with onset on or after the first dose and up to the end of the study (week 36).
Arm/Group | Verinurad + Allopurinol | Allopurinol | Placebo
All-Cause Mortality (participants affected / at risk) | 1/53 | 2/53 | 1/53
Serious Adverse Events (participants affected / at risk) | 10/53 | 10/53 | 9/53
Other Adverse Events (participants affected / at risk) | 24/53 | 26/53 | 20/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verinurad + Allopurinol (N=53) | Allopurinol (N=53) | Placebo (N=53)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fissure haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 5 (8) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verinurad + Allopurinol (N=53) | Allopurinol (N=53) | Placebo (N=53)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 3 (4) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 2 (3)
Cardiac failure (Cardiac disorders) | 4 (7) | 1 (1) | 4 (5)
Blood creatinine increased (Investigations) | 2 (2) | 5 (5) | 2 (2)
Blood pressure increased (Investigations) | 3 (3) | 1 (1) | 2 (2)
Weight increased (Investigations) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT04327024/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT04327024/SAP_001.pdf